CLINICAL TRIAL: NCT06544902
Title: Virtual Reality Intervention for Stress, Resilience, and Blood Pressure Management in Black Women
Brief Title: Virtual Reality Intervention for Stress, Resilience, and Blood Pressure Management in Black Women - Realist Women Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Judite Blanc, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240402; 1K01HL175286-01 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Stress; Hypertension
Keywords: Intersectional Framework
MeSH Terms: conditions — Hypertension; Intersectional Framework

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-Stress Management Group (Experimental): Participants in this group will receive VR intervention for up to 6 months
  Interventions: Other: VR Stress Management
- Education Control Group (Active Comparator): Participants in this group will be exposed to standard care through educational materials for up to 6 months.
  Interventions: Behavioral: Education Control

INTERVENTIONS:
Other: VR Stress Management — First Resort (FR) is an eight-week wellness program that comprises 22 modules, each lasting between 10 and 20 minutes, participants will complete modules weekly in person. Each module will teach participants about values-based goal setting/ behavioral activation, and cognitive restructuring.
  Arms: VR-Stress Management Group
Behavioral: Education Control — Participants in this group will receive one-time educational material regarding stress. The participants can review the material remotely. American Heart Association (AHA) brochures and infographics regarding chronic stress and women's health, heart disease and mental health among black women, healthy for good sleep well, among other useful resources.
  Arms: Education Control Group

SUMMARY:
The Realist Women Study wants to see if a special program using virtual reality can help Black women deal with stress and improve Black women's heart health. The study team wants to see if using virtual reality (VR) can help with stress of Black women. The investigator will look at things like sleep, stress, and how well the VR works. The investigator also wants to know about any problems Black women might have using virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as a Black woman
* at least 21 years of age
* fluency in English
* International Classification of Diseases (ICD)10 diagnosis of hypertension
* being a South Florida resident
* willing to be audio-recorded

Exclusion Criteria:

* History of psychosis disorders
* absence of vision and cognitive impairment
* absence of epilepsy disorders
* absence of motion sickness.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in stress as measured by Perceived Stress Scale (PSS) | Baseline and up to 6 months
  scores ranging from 0 (no symptoms) to 40 (highest severity).
Change in discrimination as measured by Intersectional Discrimination Index (InDI) | Baseline and up to 6 months
  scores ranging from 0 to 4; higher scores indicate greater anticipated intersectional discrimination.
Change in Traumatic stress as measured by Life Events Checklist | Baseline and up to 6 months
  This self-report checklist screens for potentially traumatic events in an individual's lifetime. Scores range from 1 to 17, higher scores indicate higher traumatic exposures. It consists of 17 questions with responses such as "happened to me," "witnessed it," "learned about it," "part of my job," "not sure," and "doesn't apply."
Change in stress as measured by the chronic stress scale | Baseline and up to 6 months
  The Chronic Stress Scale is a 51-item scale that evaluates the perceived experience of chronic stress. Scores range from 0 (not true) to 2 (very true).
Change in stress as measured by the Stress in Context (SIC) Questionnaire | Baseline and up to 6 months
  The SIC Questionnaire is a 21-item survey assessing stress perception in specific contexts (e.g., home, work, social relationships), with scoring from 1 (never) to 4 (usually).
Change in stress as measured by the Giscombe Superwoman Schema Questionnaire | Baseline and up to 6 months
  It contains 35 statements rated from 0 (not true) to 4 (true all the time) across the 5 subscales. subscale items are summed to create one Super Woman Schema (SWS) total, these categories can be used: 0-35: Low SWS 36-70: Moderate SWS 71-105: High SWS

SECONDARY OUTCOMES:
Change in resiliency as measured by Connor-Davidson Resilience Scale (CD-RISC) | Baseline and up to 6 months
  Scores range from 0-40 higher scores indicate higher resiliency
Change in objective sleep health as measured by Sleep Health Objective | Baseline and up to 6 months
  Sleep will be assessed using actigraphy measured in hours.
Change in blood pressure | Baseline and up to 3 months after intervention
  Measured by millimeter of mercury

CONTACTS AND LOCATIONS:
Overall Officials: Judite Blanc, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No